CLINICAL TRIAL: NCT01571635
Title: A Phase 2A, Open-label Dose Finding Study to Determine the Safety and Tolerability of Sotatercept (ACE-011) in Adults With BETA(b)-THALASSEMIA.
Brief Title: Study to Determine the Safety and Tolerability of Sotatercept (ACE-011) in Adults With Beta( β)- Thalassemia.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-011-B-THAL-001; 2011-005659-15 (EudraCT Number)
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Beta Thalassemia Major; Beta Thalassemia Intermedia
Keywords: Beta-Thalassaemia
MeSH Terms: conditions — beta-Thalassemia | interventions — ACE-011

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sotatercept dose level 0.1mg/kg (Experimental): Experimental 0.1 mg/kg -Sotatercept will be administered as a subcutaneous injection once every 21 days during the treatment period
  Interventions: Drug: SOTATERCEPT (ACE-011)
- Sotatercept dose level 0.3mg/ kg (Experimental): Experimental 0.3 mg/kg - Sotatercept will be administered as a subcutaneous injection once every 21 days during the treatment period
  Interventions: Drug: SOTATERCEPT (ACE-011)
- Sotatercept dose level 0.5mg/kg (Experimental): Experimental 0.5 mg/kg -Sotatercept will be administered as a subcutaneous injection once every 21 days during the treatment period
  Interventions: Drug: SOTATERCEPT (ACE-011)
- Sotatercept dose level 0.75mg/kg (Experimental): Experimental 0.75 mg/kg - Sotatercept will be administered as a subcutaneous injection once every 21 days during the treatment period
  Interventions: Drug: SOTATERCEPT (ACE-011)
- Sotatercept dose level 1.0mg/kg (Experimental): Experimental 1.0 mg/kg -Sotatercept will be administered as a subcutaneous injection once every 21 days during the treatment period
  Interventions: Drug: SOTATERCEPT (ACE-011)
- Sotatercept dose level 1.5mg/kg (Experimental): Experimental 1.5 mg/kg -Sotatercept will be administered as a subcutaneous injection once every 21 days during the treatment period
  Interventions: Drug: SOTATERCEPT (ACE-011)

INTERVENTIONS:
Drug: SOTATERCEPT (ACE-011) — 0.1 mg/kg to 1.5mg/kg Sotatercept will be administered as a subcutaneous injection once every 21 days during the treatment period.
  Other Names: (ACE-011)

SUMMARY:
Dose finding study to determine the safety and tolerability of Sotatercept (ACE-011) in adults with Beta (β)-Thalassemia

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age at the time of signing the informed consent document with a diagnosis of β-thalassemia major (including all subtypes) or β-thalassemia intermedia.
* For transfusion dependent subjects: permanent transfusion dependency is defined as requiring packed red blood cells (pRBCs) and iron chelation therapy:

  * Average transfusion requirement of at least 2 units/30 days of pRBCs (Gale, 2011) confirmed for a minimum of 168 days (six months) immediately preceding enrollment (study Day 1, first Dose);
  * No transfusion-free period of more than 45 consecutive days during the 168 days immediately preceding enrollment (study Day 1, first Dose);
  * Prior transfusion hemoglobin levels ≤ 10.5 g/dL.
* For non-transfusion dependent subjects: non-transfusion dependency is defined as a transfusion free for a minimum of 168 days immediately preceding enrollment (study Day 1, first Dose), with the exception of ≤ to one episode of transfusion in the period of a minimum of 168 days immediately preceding enrollment (study Day 1, first Dose) (One episode of transfusion is defined as ≤ 4 transfusion units administered, occurred within 42 days [first transfusion is counted as day 1] due to concurrent illness [e.g. infection], [Guidelines Clin Management of Thalassaemia, 2008]). (This inclusion criteria is not valid for France).
* Performance status: Eastern Cooperative Oncology Group (ECOG) score of 0 to 1
* No concurrent severe hepatic disease:

  * Aspartate Aminotransferase (AST) or Alanine Transaminase (ALT) no greater than 3 x upper limit of normal (ULN);
  * Albumin ≥ 3 g/dL.
* Serum creatinine ≤ 1.5 x ULN.
* Females of childbearing potential participating in the study are to use highly effective methods of birth control during study participation and for 112 days (approximately five times the mean terminal half-life of sotatercept [23 days] based on multiple-dose PK data) following the last dose of sotatercept. FCBP must have a negative serum beta Human Chorionic Gonadotropin (β-HCG) pregnancy test within three days of Sotatercept dosing (Day 1). Subjects must be counseled concerning measures to be used to prevent pregnancy and potential toxicities prior to the first dose of sotatercept. A FCBP is a sexually mature woman who has not undergone a hysterectomy or bilateral oophorectomy or who has not been postmenopausal for at least 24 consecutive months (i.e., who has had menses at some time in the preceding 24 months).
* Males must agree to use a latex condom during any sexual contact with FCBSs while participating in the study and for 112 days following the last dose of Sotatercept, even if he has undergone a successful vasectomy. Subjects must be counseled concerning measures to be used to prevent pregnancy and potential toxicities prior to the first dose of sotatercept.
* Agreement to adhere to the study visit schedule, understand and comply with all protocol requirements.
* Understand and provide written informed consent.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing participating in the study.
* Evidence of active Hepatitis C antibody (HCV), Hepatitis B surface antigen (HBsAg and HB core Ab), or Human Immunodeficiency Virus (HIV) antibody.
* Known history of thromboembolic events ≥ Grade 3 according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 (current active minor version).
* Subjects with insulin dependent diabetes.
* Subjects with major cardiac problems such as:

  * Major risk of heart failure, confirmed with myocardiac T2* ≤ 10 ms. Myocardiac T2* performed in the last one and a half years prior to subject enrollment (study Day 1, first Dose) will be considered valid.
  * Cardiac arrhythmia which requires treatment (i.e. atrial fibrillation).
* Treatment with another investigational drug or device < 28 days prior to study entry.
* Use of an Erythropoiesis Stimulating Agent (ESA) within the 28 days prior to enrollment (study Day 1, first Dose).
* Subjects on hydroxyurea treatment for which the dose was changed in the last one year prior to subject enrollment (study Day 1, first Dose).
* Subjects on anticoagulant therapy, such as warfarin.
* Subjects who started bisphosphonates within the last three months prior to subject enrollment (study Day 1, first Dose).
* Pregnant or lactating females.
* Uncontrolled hypertension. Controlled hypertension for this protocol is considered ≤ Grade 1 according to NCI CTCAE version 4.0 (current active minor version) (Appendix B).
* A history of major organ damage including:

  * Liver disease with ALT > 3x ULN or histopathological evidence of liver cirrhosis on liver biopsy;
  * Heart disease with ejection fraction ≥ Grade 2 according to NCI CTCAE version 4.0 (current active minor version);
  * Kidney disease with a calculated creatinine clearance < 40 mL/min (Cockcroft-Gault formula);
  * Pulmonary fibrosis or pulmonary hypertension as confirmed by a specialist.
* Adrenal insufficiency.
* Heart failure as classified by the New York Heart Association (NYHA) classification of 3 or higher (Appendix C).
* Major surgery within 30 days prior to study Day 1 (subjects must have completely recovered from any previous surgery prior to study Day 1).
* History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the Investigational Product (see Investigator Brochure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-10-10 (Actual); Primary Completion 2015-07-02 (Actual); Study Completion 2022-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (18):
- France (5):
  - Hopital Henri Mondor, Créteil
  - Groupe Hospitalier Henri Mondor, Créteil
  - Hospital of Necker, Paris
  - Local Institution - 001, Paris
  - Hôpital Necker-Enfants Malades, Paris
- Greece (2):
  - Local Institution - 300, Ampelokipi - Athens
  - Laiko General Hospital, Ampelokipi - Athens
- Italy (8):
  - Universita degli Studi di Cagliari - ASL8, Cagliari
  - Universita Degli Studi Di Cagliari, Cagliari
  - Local Institution - 200, Genoa
  - Ospedale Galliera, Genoa
  - Ente Ospedaliero Ospedali Galliera, Genova
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS Ospedale Maggiore, Milan
  - Local Institution - 201, Milan
- United Kingdom (3):
  - Local Institution - 100, London
  - UCL Cancer Institute, London
  - UCL Cancer Institue, London

REFERENCES:
- [Background] Cappellini MD, Porter J, Origa R, Forni GL, Voskaridou E, Galacteros F, Taher AT, Arlet JB, Ribeil JA, Garbowski M, Graziadei G, Brouzes C, Semeraro M, Laadem A, Miteva D, Zou J, Sung V, Zinger T, Attie KM, Hermine O. Sotatercept, a novel transforming growth factor beta ligand trap, improves anemia in beta-thalassemia: a phase II, open-label, dose-finding study. Haematologica. 2019 Mar;104(3):477-484. doi: 10.3324/haematol.2018.198887. Epub 2018 Oct 18. PMID 30337358
- [Background] Cappellini M, et al. A Phase 2a, Open-Label, Dose-Finding Study to Determine the Safety and Tolerability of Sotatercept (ACE-011) in Adults With Beta ( )-Thalassemia: Interim Results. Presented at the 55th Annual Meeting of the American Society of Hematology (ASH), December 7-10, 2013, New Orleans, LA. Abstract No. 3448
- [Background] "Porter J, et al. Interim Results From a Phase 2A, Open-Label, Dose-Finding Study To Determine The Safety, Efficacy, And Tolerability of Sotatercept (ACE-001) In Adults with Beta-Thalassemia. Presented at the 19thCongress of the European Hematology Association, June 12-15, 2015, Milan, Italy. Abstract No. S622 "
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/us/en/home.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Sponsor decided to stop advancing sotatercept development in the β-thalassemia indication; therefore, the study participants enrollment stopped during the Treatment Period. No participants were enrolled in the dose level 1.5 mg/kg that was planned in the protocol.
  Additionally, the protocol planned to enroll approximately 30 participants in an expansion cohort once the potential recommended dose (PRD) was defined. Due to early termination of the study, the expansion cohort was not opened.
Groups:
- Dose Level 1a: 0.1 mg/kg: Dose level 1a (starting dose) 0.1 mg/kg Sotatercept will be administered as an SC injection once every 21 days for up to six planned doses during the Treatment Period.
- Dose Level 1b: 0.3 mg/kg: Dose level 1b (starting dose) 0.3 mg/kg Sotatercept will be administered as an SC injection once every 21 days for up to six planned doses during the Treatment Period.
- Dose Level 2: 0.5 mg/kg: Dose level 2 (escalation dose) 0.5 mg/kg Sotatercept will be administered as an SC injection once every 21 days for up to six planned doses during the Treatment Period.
- Dose Level 3: 0.75 mg/kg: Dose level 3 (escalation dose) 0.75 mg/kg Sotatercept will be administered as an SC injection once every 21 days for up to six planned doses during the Treatment Period.
- Dose Level 4: 1 mg/kg: Dose level 4 (escalation dose) 1 mg/kg Sotatercept will be administered as an SC injection once every 21 days for up to six planned doses during the Treatment Period.
Period: Overall Study
Arm/Group | Dose Level 1a: 0.1 mg/kg | Dose Level 1b: 0.3 mg/kg | Dose Level 2: 0.5 mg/kg | Dose Level 3: 0.75 mg/kg | Dose Level 4: 1 mg/kg
Started | 8 | 9 | 8 | 12 | 9
Completed | 2 | 1 | 1 | 0 | 0
Not Completed | 6 | 8 | 7 | 12 | 9
Not completed — Adverse Event | 3 | 0 | 2 | 3 | 5
Not completed — Other reasons | 2 | 1 | 2 | 2 | 1
Not completed — Study terminated by sponsor | 0 | 4 | 1 | 3 | 1
Not completed — Withdrew consent | 1 | 1 | 2 | 3 | 0
Not completed — Lack of Efficacy | 0 | 2 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1a: 0.1 mg/kg | Dose Level 1b: 0.3 mg/kg | Dose Level 2: 0.5 mg/kg | Dose Level 3: 0.75 mg/kg | Dose Level 4: 1 mg/kg | Total
Number analyzed (Participants) | 8 | 9 | 8 | 12 | 9 | 46
Age, Continuous [Median (Standard Deviation); unit: Years] | 39.5 (8.21) | 40.0 (9.89) | 38.5 (7.63) | 44.0 (10.29) | 41.0 (10.36) | 39.5 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 8 | 3 | 22
  Male | 4 | 5 | 5 | 4 | 6 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 7 | 9 | 6 | 10 | 8 | 40
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Potential Recommended Dose as Determined by Number of Participants Experiencing Dose-Limiting Toxicities and Recommended Dose
Description: Number of participants with dose-limiting toxicities (DLT) are used to determine the potential recommended dose (PRD). PRD is defined as the highest dose with up to 1 out of 6 patients experiencing a DLT. DLT is defined as any side effects of the study treatment serious enough to prevent an increase in dose or level of treatment, including at least one of the following: Hypertension ≥ Grade 3 per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0; Hgb > 14 g/dL sustained for four weeks; any NCI CTCAE toxicity ≥ Grade 3. Grade 3 is defined as severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily life.
  PRD was identified as 1 mg/kg. Due to study termination, no patients were enrolled after 1 mg/kg cohort or in the Expansion Cohort. Thus, primary analyses to determine recommended dose (RD) were not conducted.
Time Frame: From first dose up to 28 days post the first dose
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1a: 0.1 mg/kg | Dose Level 1b: 0.3 mg/kg | Dose Level 2: 0.5 mg/kg | Dose Level 3: 0.75 mg/kg | Dose Level 4: 1 mg/kg
Number analyzed (Participants) | 8 | 9 | 8 | 12 | 9
Participants | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Red Blood Cell Transfusion Burden Reduction From Baseline During Treatment
Description: Transfusion burden at baseline is defined as the total number of units of RBC transfusions that participants received within 168 days (24 weeks) prior to the first dose of study therapy. Transfusion burden during treatment is defined as the total number of RBC transfusion units that each participant received during the treatment divided by the treatment duration and multiplied by 168 days. The result is a 168-day transfusion burden average. Baseline measurement includes RBC transfusion history for transfusion dependent and non-transfusion dependent participants, starting at 168 days prior to enrollment.
Time Frame: From baseline to the last dose of study treatment (up to approximately 112 months)
Population: Safety Population Transfusion Dependent-All participants who received at least one dose of sotatercept and are transfusion dependent.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1a: 0.1 mg/kg | Dose Level 1b: 0.3 mg/kg | Dose Level 2: 0.5 mg/kg | Dose Level 3: 0.75 mg/kg | Dose Level 4: 1 mg/kg
Number analyzed (Participants) | 2 | 3 | 2 | 5 | 4
Participants
  ≥ 25% reduction | 0 | 0 | 2 | 4 | 3
  ≥ 33% reduction | 0 | 0 | 2 | 3 | 1
  ≥ 50% reduction | 0 | 0 | 1 | 2 | 0

3. Secondary Outcome: Number of Participants With Hemoglobin Level Increase From Baseline in Non-Transfusion Dependent B-Thalassemia Intermedia Participants
Description: The Number of participants with a change in Hemoglobin levels will be listed for non-RBC transfusion dependent participants. Baseline assessments are the average of the last two measurements prior to the start of therapy.
Time Frame: Measurements were taken in 9 and 12-week intervals, from baseline up to approximately 112 months
Population: Non-RBC transfusion dependent participants-participants who are in the safety population and are not transfusion dependent. This is a subgroup of the B-thalassemia intermedia population.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1a: 0.1 mg/kg | Dose Level 1b: 0.3 mg/kg | Dose Level 2: 0.5 mg/kg | Dose Level 3: 0.75 mg/kg | Dose Level 4: 1 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 5
Participants
  9-week episode with Hgb ≥ 1.0 g/dl change from baseline (non-transfusion dependent participants) | 0 | 5 | 4 | 6 | 2
  9-week episode with Hgb ≥ 1.5 g/dl change from baseline (non-transfusion dependent participants) | 0 | 2 | 2 | 6 | 1
  12-Week episode with Hgb ≥ 1.0 g/dl change from baseline (non-transfusion dependent participants) | 0 | 4 | 4 | 6 | 1
  12-Week episode with Hgb ≥ 1.5 g/dl change from baseline (non-transfusion dependent participants) | 0 | 2 | 2 | 6 | 1

4. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Adverse events are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal. Treatment emergent adverse events (TEAE) are defined as an AE that began after the start of trial medication treatment; or if the event was continuous from baseline and was serious, trial medication-related, or resulted in death, discontinuation, or interruption or reduction of trial therapy.
Time Frame: From first dose up to 112 days after the last dose of study treatment (up to 115 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1a: 0.1 mg/kg | Dose Level 1b: 0.3 mg/kg | Dose Level 2: 0.5 mg/kg | Dose Level 3: 0.75 mg/kg | Dose Level 4: 1 mg/kg
Number analyzed (Participants) | 8 | 9 | 8 | 12 | 9
Participants
  Participants with at least one TEAE | 8 | 9 | 8 | 12 | 9
  TEAE leading to dose interruption | 2 | 5 | 4 | 2 | 5
  Participants with at least one serious TEAE | 3 | 3 | 3 | 3 | 3
  Participants with at least one grade 2/3/4 TEAE | 7 | 9 | 6 | 11 | 9
  Participants with at least one drug-related grade 2/3/4 TEAE | 4 | 3 | 4 | 7 | 7
  Participants with at least one serious drug- related TEAE | 2 | 1 | 1 | 0 | 1
  Participants with at least one TEAE leading to sotatercept withdrawal | 3 | 0 | 2 | 3 | 5

5. Secondary Outcome: Concentrations of Sotatercept in Serum
Description: Sotatercept was administered as a subcutaneous injection every 21 days during the Treatment Period. Pharmacokinetic (PK) samples were collected at the pre-specified timepoints.
Time Frame: Dose 1, Day 8; Dose 1, Day 15; Dose 2, Day 1; Dose 2, Day 8; Dose 3, Day 1; Dose 3, Day 8; Dose 4, Day 1; Dose 5, Day 1; Dose 6, Day 1
Population: All treated participants
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Dose Level 1a: 0.1 mg/kg | Dose Level 1b: 0.3 mg/kg | Dose Level 2: 0.5 mg/kg | Dose Level 3: 0.75 mg/kg | Dose Level 4: 1 mg/kg
Number analyzed (Participants) | 8 | 9 | 8 | 12 | 9
ng/mL
  Dose 1, Day 8: number analyzed (Participants) | 8 | 8 | 8 | 12 | 9
  Dose 1, Day 8 | 598.3 [289.2 to 1345.4] | 1454.05 [1006.6 to 2768.3] | 3045.45 [1586.7 to 4480] | 5837.65 [3238.1 to 10590.5] | 3874 [2264.9 to 7003]
  Dose 1, Day 15 | 388.7 [98.4 to 1046] | 1150.1 [550.3 to 2158.4] | 2329.75 [952 to 3005.5] | 4279.65 [2107.8 to 6692] | 2405.6 [1825.3 to 4605.5]
  Dose 2, Day 1 | 294.75 [112.9 to 547.1] | 770.3 [317.2 to 1300.1] | 1468.05 [682 to 2550.5] | 2955.2 [1257.5 to 4450.8] | 1701.5 [888.6 to 4267.9]
  Dose 2, Day 8 | 683.1 [250.1 to 1210.6] | 2065 [1363.7 to 3626.4] | 4136.8 [1661.9 to 5573.8] | 7753.35 [5046.4 to 8805.6] | 5148.1 [3537.4 to 10418.7]
  Dose 3, Day 1 | 325.35 [228.8 to 790] | 956.8 [380.6 to 1552.6] | 2157.3 [422 to 3088.4] | 3628.45 [653.5 to 6429.1] | 2602.6 [822.2 to 5668.1]
  Dose 3, Day 8: number analyzed (Participants) | 6 | 9 | 7 | 12 | 7
  Dose 3, Day 8 | 758.1 [444 to 1232] | 2319.9 [1475.6 to 3667.4] | 4507.3 [2077.8 to 5762.3] | 8373.05 [5345.5 to 12177.8] | 6050.8 [3892.5 to 12139.6]
  Dose 4, Day 1: number analyzed (Participants) | 6 | 9 | 7 | 11 | 8
  Dose 4, Day 1 | 334.85 [298 to 1014.9] | 1022.3 [348.8 to 2096.9] | 2441.6 [784 to 2845.3] | 4137.1 [1447.1 to 6126.6] | 2869.2 [1478.9 to 4787.7]
  Dose 5, Day 1: number analyzed (Participants) | 4 | 6 | 7 | 9 | 8
  Dose 5, Day 1 | 385.1 [287.5 to 467.5] | 1473.9 [762.1 to 2764.4] | 1618.8 [953.4 to 3440] | 4449.7 [2340.4 to 5887.8] | 3048 [1125.5 to 6529.3]
  Dose 6, Day 1: number analyzed (Participants) | 4 | 8 | 5 | 10 | 8
  Dose 6, Day 1 | 297.60 [227.80 to 484.40] | 1368.10 [449.70 to 2363.20] | 2266.40 [1115.20 to 3788.50] | 4062.80 [1481.10 to 6584.00] | 2780.80 [1479.20 to 7896.70]

6. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA)
Description: The number of participants with Anti-Sotatercept Antibody is a summary of antidrug antibody (ADA) status for ADA-evaluated participants. A participant is counted as 'positive' if there is any positive result captured during the study, a participant is counted as 'negative' if there is no positive result captured during the study. ADA data was collected Day 1 in dose schedules 1 through 6. Starting from Dose 7, ADA was measured at Day 1 every 3 Doses, then finally at the post-treatment follow-up visit at Month 2 and Month 4.
Time Frame: From first dose up to 4 months after last dose (up to approximately 116 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1a: 0.1 mg/kg | Dose Level 1b: 0.3 mg/kg | Dose Level 2: 0.5 mg/kg | Dose Level 3: 0.75 mg/kg | Dose Level 4: 1 mg/kg
Number analyzed (Participants) | 8 | 9 | 8 | 12 | 9
Participants
  Negative | 8 | 8 | 8 | 10 | 9
  Positive | 0 | 1 | 0 | 2 | 0

7. Secondary Outcome: Number of Participants Experiencing Quality of Life (QOL) Change From Baseline
Description: The number of participants in the expansion cohort experiencing changes from baseline in Quality of Life. QOL was planned to be assessed at Day 168 (6 months) and Day 336 (12 months), after Dose 1 Day 1, independent of Dose Delay for participants enrolled in the Expansion Cohort only. QOL was planned to be calculated using the SF-36 and the FACT Anemia. The SF-36 is a Medical Outcomes Study (MOS) consisting of 36 questions developed to determine health status. The SF-36 measures eight scales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The FACT Anemia measures fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) Measurement System.
  Due to early study termination, no participants were enrolled in the expansion cohort and QOL was not assessed.
Time Frame: From pre-dose up to Dose 8 (168 days/6months) and Dose 16 (336 days/12months) only
Population: Expansion cohort
Arm/Group | Dose Level 1a: 0.1 mg/kg | Dose Level 1b: 0.3 mg/kg | Dose Level 2: 0.5 mg/kg | Dose Level 3: 0.75 mg/kg | Dose Level 4: 1 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their enrollment to study completion, (up to approximately 115 months). SAEs and Other AEs were assessed from first dose to 112 days following last dose (up to approximately 115 months)
Arm/Group | Dose Level 1a: 0.1 mg/kg | Dose Level 1b: 0.3 mg/kg | Dose Level 2: 0.5 mg/kg | Dose Level 3: 0.75 mg/kg | Dose Level 4: 1 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/8 | 0/12 | 0/9
Serious Adverse Events (participants affected / at risk) | 3/8 | 3/9 | 3/8 | 3/12 | 3/9
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9 | 8/8 | 12/12 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1a: 0.1 mg/kg (N=8) | Dose Level 1b: 0.3 mg/kg (N=9) | Dose Level 2: 0.5 mg/kg (N=8) | Dose Level 3: 0.75 mg/kg (N=12) | Dose Level 4: 1 mg/kg (N=9)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
EXTRAMEDULLARY HAEMOPOIESIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
SUBILEUS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
FATIGUE (General disorders) | 0 | 0 | 1 | 0 | 0
LOCAL SWELLING (General disorders) | 0 | 0 | 1 | 0 | 0
PYREXIA (General disorders) | 0 | 1 | 1 | 0 | 0
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 0 | 1 | 0 | 0
BACTERIAL PROSTATITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
CORONA VIRUS INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0
PHARYNGOTONSILLITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
ULNA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 1 | 0 | 0 | 0 | 0
THROMBOSIS (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1a: 0.1 mg/kg (N=8) | Dose Level 1b: 0.3 mg/kg (N=9) | Dose Level 2: 0.5 mg/kg (N=8) | Dose Level 3: 0.75 mg/kg (N=12) | Dose Level 4: 1 mg/kg (N=9)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
BONE MARROW OEDEMA SYNDROME (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
EXTRAMEDULLARY HAEMOPOIESIS (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 2
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2 | 0
SPLENOMEGALY (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
EXTRASYSTOLES (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
LEFT ATRIAL DILATATION (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
PALPITATIONS (Cardiac disorders) | 0 | 2 | 0 | 0 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
SPLINTER HAEMORRHAGES (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
TACHYCARDIA (Cardiac disorders) | 0 | 2 | 0 | 1 | 1
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
BENIGN FAMILIAL HAEMATURIA (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
DEAFNESS (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
EAR PAIN (Ear and labyrinth disorders) | 0 | 1 | 1 | 2 | 1
EXTERNAL EAR INFLAMMATION (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
TINNITUS (Ear and labyrinth disorders) | 0 | 2 | 0 | 1 | 2
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0
AUTOIMMUNE THYROIDITIS (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
HYPERPROLACTINAEMIA (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
HYPERTHYROIDISM (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
THYROID CYST (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
THYROIDITIS (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
BLEPHARITIS (Eye disorders) | 0 | 0 | 0 | 0 | 1
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 | 0 | 0 | 0 | 1
CONJUNCTIVITIS (Eye disorders) | 0 | 1 | 1 | 1 | 1
CONJUNCTIVITIS ALLERGIC (Eye disorders) | 0 | 0 | 0 | 0 | 1
DACRYOSTENOSIS ACQUIRED (Eye disorders) | 0 | 1 | 0 | 0 | 0
EYE PAIN (Eye disorders) | 0 | 1 | 0 | 0 | 0
EYE SWELLING (Eye disorders) | 0 | 1 | 0 | 1 | 0
LACRIMAL DISORDER (Eye disorders) | 0 | 1 | 0 | 0 | 0
LACRIMATION INCREASED (Eye disorders) | 0 | 0 | 0 | 1 | 0
OCULAR HYPERAEMIA (Eye disorders) | 0 | 0 | 0 | 1 | 0
PINGUECULA (Eye disorders) | 0 | 0 | 1 | 0 | 0
PTERYGIUM (Eye disorders) | 0 | 0 | 0 | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 3 | 3 | 1 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 5 | 1 | 4 | 1
ANAL PRURITUS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
COLITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 3 | 0 | 2 | 1
DENTAL CARIES (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
DENTAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 4 | 1 | 2 | 1
DUODENOGASTRIC REFLUX (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 2
FAECALOMA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
FOOD POISONING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
HYPERCHLORHYDRIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
LIP DISCOLOURATION (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
MOUTH ULCERATION (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 3 | 4 | 3 | 1
ODYNOPHAGIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
ORAL DISORDER (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
PARAESTHESIA ORAL (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
PAROTID GLAND ENLARGEMENT (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
TEETHING (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 0
TOOTHACHE (Gastrointestinal disorders) | 1 | 4 | 3 | 1 | 1
VOMITING (Gastrointestinal disorders) | 1 | 2 | 2 | 2 | 0
ASTHENIA (General disorders) | 4 | 4 | 4 | 5 | 3
CHEST DISCOMFORT (General disorders) | 0 | 1 | 1 | 0 | 0
CHEST PAIN (General disorders) | 0 | 1 | 0 | 0 | 0
CHILLS (General disorders) | 0 | 0 | 0 | 1 | 0
CYST (General disorders) | 1 | 0 | 0 | 0 | 0
FATIGUE (General disorders) | 0 | 1 | 4 | 2 | 2
GENERALISED OEDEMA (General disorders) | 0 | 0 | 1 | 0 | 0
GRANULOMA (General disorders) | 0 | 1 | 0 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 4 | 3 | 1 | 0
INJECTION SITE ERYTHEMA (General disorders) | 0 | 0 | 0 | 1 | 0
INJECTION SITE INFLAMMATION (General disorders) | 0 | 0 | 0 | 0 | 1
IRRITABILITY (General disorders) | 0 | 0 | 0 | 1 | 0
LOCAL SWELLING (General disorders) | 1 | 2 | 1 | 1 | 0
LOCALISED OEDEMA (General disorders) | 0 | 1 | 0 | 0 | 0
MALAISE (General disorders) | 0 | 1 | 1 | 0 | 0
MUCOSAL HYPERAEMIA (General disorders) | 0 | 0 | 1 | 0 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 1 | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 2 | 0 | 1 | 0 | 1
PAIN (General disorders) | 0 | 0 | 2 | 1 | 0
PYREXIA (General disorders) | 3 | 6 | 2 | 3 | 4
VACCINATION SITE ERYTHEMA (General disorders) | 0 | 1 | 0 | 0 | 0
VACCINATION SITE LYMPHADENOPATHY (General disorders) | 0 | 0 | 0 | 0 | 1
VACCINATION SITE PAIN (General disorders) | 0 | 2 | 0 | 0 | 0
VACCINATION SITE SWELLING (General disorders) | 0 | 1 | 0 | 0 | 0
VACCINATION SITE WARMTH (General disorders) | 0 | 1 | 0 | 0 | 0
DEFICIT FOLATE (General disorders) | 1 | 0 | 0 | 0 | 0
BILIARY DILATATION (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
CHOLESTASIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
GALLBLADDER POLYP (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
HEPATOCELLULAR INJURY (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
PORTAL HYPERTENSION (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
ALLERGY TO ARTHROPOD STING (Immune system disorders) | 0 | 0 | 1 | 0 | 0
ALLOIMMUNISATION (Immune system disorders) | 0 | 0 | 0 | 0 | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 0 | 1 | 0 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 0 | 0 | 1
HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 1 | 1 | 1
SEASONAL ALLERGY (Immune system disorders) | 0 | 1 | 1 | 0 | 1
ACNE PUSTULAR (Infections and infestations) | 0 | 0 | 0 | 1 | 0
ACUTE SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
ACUTE TONSILLITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
BODY TINEA (Infections and infestations) | 0 | 0 | 1 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 4 | 1 | 1 | 1
CONJUNCTIVITIS VIRAL (Infections and infestations) | 0 | 0 | 0 | 1 | 0
CYSTITIS (Infections and infestations) | 1 | 0 | 1 | 2 | 0
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1
EAR INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 2
EYE INFECTION (Infections and infestations) | 0 | 0 | 1 | 1 | 0
EYELID INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1
FOLLICULITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 1 | 1 | 0 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 1 | 0 | 1 | 1
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
GINGIVAL INFECTION (Infections and infestations) | 0 | 2 | 0 | 0 | 0
GINGIVITIS (Infections and infestations) | 0 | 2 | 1 | 0 | 0
HELICOBACTER INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 1
HORDEOLUM (Infections and infestations) | 0 | 0 | 1 | 0 | 1
INFECTED BITES (Infections and infestations) | 0 | 1 | 0 | 1 | 0
INFECTED SKIN ULCER (Infections and infestations) | 0 | 0 | 1 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 5 | 1 | 1 | 1
KLEBSIELLA INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 2 | 1 | 1 | 1
NASOPHARYNGITIS (Infections and infestations) | 2 | 1 | 4 | 1 | 2
ONYCHOMYCOSIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ORAL HERPES (Infections and infestations) | 2 | 4 | 0 | 0 | 1
OTITIS EXTERNA (Infections and infestations) | 0 | 0 | 1 | 0 | 0
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0
PARONYCHIA (Infections and infestations) | 0 | 0 | 1 | 0 | 0
PERIODONTITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0
PHARYNGITIS (Infections and infestations) | 1 | 2 | 0 | 1 | 2
PNEUMONIA VIRAL (Infections and infestations) | 0 | 0 | 0 | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 | 0 | 0 | 0 | 1
RHINITIS (Infections and infestations) | 1 | 3 | 5 | 1 | 1
SINUSITIS (Infections and infestations) | 0 | 2 | 2 | 0 | 1
TINEA PEDIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0
TONSILLITIS (Infections and infestations) | 0 | 1 | 0 | 1 | 1
TOOTH ABSCESS (Infections and infestations) | 0 | 2 | 0 | 0 | 2
TOOTH INFECTION (Infections and infestations) | 0 | 1 | 2 | 0 | 0
TRACHEITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
TROPICAL ULCER (Infections and infestations) | 0 | 0 | 1 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 2 | 4 | 1 | 2
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 2 | 1 | 1
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 | 0 | 1 | 0 | 0
URINARY TRACT INFECTION FUNGAL (Infections and infestations) | 0 | 0 | 0 | 1 | 0
VAGINAL INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 1 | 0
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
ARTHROPOD STING (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
CHEST INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0 | 0
EPICONDYLITIS (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
HAEMOLYTIC TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
LACERATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 2
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
MENISCUS INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
NAIL INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0 | 0
REPETITIVE STRAIN INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
TOOTH INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
VACCINATION COMPLICATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 1 | 1 | 1 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1 | 0 | 1 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0
BLOOD FOLATE DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0
BLOOD FOLLICLE STIMULATING HORMONE DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 | 0 | 0 | 1 | 1
BLOOD PRESSURE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1
CARDIAC INDEX INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0
CULTURE STOOL POSITIVE (Investigations) | 0 | 0 | 0 | 1 | 0
EJECTION FRACTION DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0
ELECTROCARDIOGRAM QT SHORTENED (Investigations) | 0 | 0 | 1 | 0 | 0
ELECTROCARDIOGRAM T WAVE ABNORMAL (Investigations) | 0 | 0 | 0 | 1 | 0
ESCHERICHIA TEST POSITIVE (Investigations) | 0 | 0 | 0 | 1 | 0
FIBRIN D DIMER INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0
GLOMERULAR FILTRATION RATE DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0
HEPATIC ENZYME INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1
PANCREATIC ENZYMES INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0
PLATELET COUNT INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0
SERUM FERRITIN INCREASED (Investigations) | 0 | 3 | 0 | 2 | 0
ULTRASOUND LIVER ABNORMAL (Investigations) | 0 | 0 | 1 | 0 | 0
ULTRASOUND SCAN ABNORMAL (Investigations) | 0 | 0 | 1 | 0 | 0
URINE PROTEIN/CREATININE RATIO INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0
VITAMIN D DECREASED (Investigations) | 0 | 1 | 0 | 0 | 0
WEIGHT DECREASED (Investigations) | 0 | 0 | 1 | 1 | 0
WEIGHT INCREASED (Investigations) | 0 | 1 | 1 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0
FOLATE DEFICIENCY (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
GOUT (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
IRON OVERLOAD (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 | 6 | 7 | 8 | 2
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 7 | 6 | 5 | 3
BONE DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 4 | 6 | 4 | 4 | 4
COCCYDYNIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
JOINT RANGE OF MOTION DECREASED (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0
LIGAMENT DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 3 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2 | 4 | 0
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4 | 2 | 2
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 5 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 3 | 5 | 5 | 3
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
SENSATION OF HEAVINESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
TEMPOROMANDIBULAR JOINT SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
TENDON PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
HAEMANGIOMA OF LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
AGEUSIA (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 3 | 3 | 3 | 2 | 0
DYSARTHRIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
DYSGEUSIA (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
FACIAL NEURALGIA (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 2 | 6 | 5 | 9 | 3
HYPERAESTHESIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
MIGRAINE (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
PRESYNCOPE (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
SCIATICA (Nervous system disorders) | 1 | 1 | 0 | 1 | 0
SINUS HEADACHE (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
SOMNOLENCE (Nervous system disorders) | 1 | 2 | 0 | 1 | 0
TREMOR (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
VISUAL FIELD DEFECT (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
ANXIETY (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0
BRUXISM (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
INSOMNIA (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
LIBIDO DECREASED (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
STRESS (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
DYSURIA (Renal and urinary disorders) | 0 | 2 | 2 | 2 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
LEUKOCYTURIA (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
MICROALBUMINURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 2
NEPHROPATHY (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 0 | 2 | 2 | 0
POLYURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
PROTEINURIA (Renal and urinary disorders) | 0 | 1 | 2 | 0 | 1
RENAL COLIC (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
RENAL CYST (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
STRANGURY (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
AMENORRHOEA (Reproductive system and breast disorders) | 1 | 2 | 0 | 2 | 0
BREAST CYST (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
CYSTOCELE (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
EPIDIDYMITIS (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
OLIGOMENORRHOEA (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 1 | 0 | 2 | 0
PELVIC PAIN (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0
PROSTATOMEGALY (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0
UTERINE PROLAPSE (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
ALLERGIC RESPIRATORY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
ASTHMATIC CRISIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 5 | 3 | 3
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 4 | 3
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
LUNG CYST (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 4 | 4 | 2
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
YAWNING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
DERMAL CYST (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
HAIR TEXTURE ABNORMAL (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
HIRSUTISM (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
PAPULE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 2 | 1
PURPURA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
SKIN HAEMORRHAGE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 0
SPIDER NAEVUS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
MENOPAUSE (Social circumstances) | 0 | 1 | 0 | 0 | 0
HAEMATOMA (Vascular disorders) | 0 | 0 | 0 | 1 | 0
HOT FLUSH (Vascular disorders) | 1 | 0 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 1 | 3 | 3 | 5 | 2
HYPOTENSION (Vascular disorders) | 2 | 1 | 2 | 0 | 0
PREHYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 1 | 0
THROMBOPHLEBITIS (Vascular disorders) | 0 | 0 | 1 | 0 | 0
VENOUS RECANALISATION (Vascular disorders) | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Sotatercept development in β-thalassemia indication was stopped and no further patients were enrolled after 1 mg/kg cohort was completed. Due to the early termination of the study and no enrollment of the Expansion Cohort, the primary analyses to determine the recommended dose (RD) and the secondary analysis of QoL change from baseline were not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.